CLINICAL TRIAL: NCT06531863
Title: A Randomized Controlled Trial to Determine the Effects of Curcumin and Epigallocatechin Gallate Supplementation on Serum Brain Derived Neurotrophic Factor and Mood Disturbance in Adults
Brief Title: Curcumin and EGCG Supplementation to Improve Serum BDNF and Mood Disturbance
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Aidan Cavanah, Graduate Assistant, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AU-STUDY00000014
Record Dates: First submitted 2024-07-16; First posted 2024-08-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-10

CONDITIONS: Mood Disturbance
MeSH Terms: interventions — Curcumin; epigallocatechin gallate

STUDY DESIGN:
Intervention Model Description: Intervention Group (supplementation with 1330mg/day curcumin and 350mg/day EGCG)
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded study with masking of participants and investigator using computer generated allocation sequences and sealed treatment and placebo supplement bags.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin and EGCG Supplementation (Experimental): Participants in the intervention group with consume 1,330mg/day curcumin with 350mg/day EGCG.
  Interventions: Dietary Supplement: Curcumin; Dietary Supplement: Epigallocatechin Gallate
- Placebo (Placebo Comparator): Participants will receive a placebo to consume everyday.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — 1,330 mg curcumin
  Arms: Curcumin and EGCG Supplementation
Dietary Supplement: Epigallocatechin Gallate — 350 mg Epigallocatechin gallate (EGCG)
  Other Names: EGCG
  Arms: Curcumin and EGCG Supplementation
Other: Placebo — Placebo to be consumed after randomization.
  Arms: Placebo

SUMMARY:
The goal of this randomized placebo controlled trial is to examine mood disturbance and serum brain derived neurotrophic factor (BDNF) in people (age 18-50) with DASS-21 subscale scores >9. The main questions it aims to answer are:

Does curcumin and EGCG supplementation improve mood disturbance symptomology? Does curcumin and EGCG supplementation increase serum BDNF? Researchers will compare intervention versus placebo.

Participants will consume an 8-week supplement of both:

* 1,330mg/day curcumin
* 350mg/day epigallocatechin gallate (EGCG)

DETAILED DESCRIPTION:
Clinical assessments will include phlebotomy (completed at weeks 0 and 8) and questionnaires which will be completed at weeks 0, 4, and 8 to assess changes in mood disorder symptomology and serum BDNF. 3 days of 24-hour diet recalls will be collected at weeks 0, 4 and 8. Daily reminders via Emitrr will be sent daily to ensure adherence to supplementation.

This is an 8-week randomized placebo controlled trial looking at mood disturbance and serum BDNF in moderately depressed adults aged 18-50. Participants will be randomized into the intervention group or placebo with the intervention group consuming 1,330mg/day curcumin and 350mg/day EGCG. Baseline mood disturbance questionnaires (DASS-21, GAD-7, GSAQ, IPAQ) and serum BDNF will be taken prior to intervention and again after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-50
* Depression subscale score of >9/21 on the DASS-21
* No change in medications or supplements over the past 3 months
* Can read and speak English

Exclusion Criteria:

* Currently consume curcumin or green tea daily
* Currently, pregnant, nursing, or trying to become pregnant
* Currently diagnosed with a perimenopausal disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in total distress as measured via DASS-21 total score. | 8-weeks
  The DASS-21 (Depression Anxiety and Stress Scale) Total ranges from 0 to 63, with lower numbers indicating less distress
Changes in serum brain derived neurotrophic factor (BDNF). | 8-weeks
  Serum BDNF will be measured via commercial ELISA kits. Higher levels of serum BDNF are optimal.

SECONDARY OUTCOMES:
Changes in DASS-21 subscales (depression, anxiety, stress). | 8-weeks
  The DASS-21 (Depression Anxiety and Stress Scale) subscales include Depression, Anxiety, and Stress, which range from 0 to 21, with lower numbers indicating less distress
Changes in subjective sleep quality. | 8-weeks
  Using Global Sleep Assessment Questionnaire includes 11 questions outlined with "During the PAST 4 WEEKS, how often" with answer choices ranging from "never, sometimes, usually and always"
Changes in subjective physical activity. | 8-weeks
  Using International Physical Activity Questionnaire has 27 questions that span 5 activity domains from "job related physical activity, transportation physical activity, house work and maintenance, recreation and sport as well as time spent sitting" over the past 7-days.
Changes in diet quality. | 8-weeks
  Using diet recalls over the past 24 hours.
Number of Participants who report daily adherence to supplementation intake | 8-weeks
  Number of participants that report consuming supplement >80% of days via daily text messages
Changes in fasting alanine aminotransferase (ALT) | 8-weeks
  Phlebotomy will be obtained while fasted 8+ hours and alanine aminotransferase (ALT) will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Changes in fasting aspartate aminotransferase (AST) | 8-weeks
  Phlebotomy will be obtained while fasted 8+ hours and aspartate transferase (AST) will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Fruge, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University School of Kinesiology, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No